CLINICAL TRIAL: NCT02452970
Title: A Phase 2, Single-Arm, Open-label, Study of RRx-001 in Second Line Treatment of Advanced Cholangiocarcinoma Prior to Readministration of First-Line Therapy
Brief Title: RRx-001 in Second Line Treatment of Advanced Cholangiocarcinoma Prior to Readministration of First-Line Therapy
Acronym: EPIC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor enrollment and adverse event experiences in the limited population
Sponsor: EpicentRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RRx001-27-01
Record Dates: First submitted 2015-05-17; First posted 2015-05-25 (Estimated); Results first posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-03

CONDITIONS: Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — RRx-001; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RRx-001 the cisplatin and gemcitabine (Experimental): Patients with advanced and metastatic biliary tract adenocarcinoma (cholangiocarcinoma) who had been treated with and failed first-line chemotherapy will be treated with RRx-001 (20 mg) intravenously weekly for up to six weeks followed by retreatment with Gemcitabine 1000 mg/m2 and Cisplatin 25 mg/m2 on Days 1 and 8 of a 21 Day Cycle until tumor progression
  Interventions: Drug: RRx-001; Drug: Gemcitabine and cisplatin

INTERVENTIONS:
Drug: RRx-001 — RRx-001 (10 mg/m2) intravenously twice weekly for up to six weeks followed by retreatment with Gemcitabine 1000 mg/m2 and Cisplatin 30 mg/m2 on Days 1 and 8 of a 21 Day Cycle until tumor progression
Drug: Gemcitabine and cisplatin — RRx-001 (20 mg) intravenously weekly for up to six weeks followed by retreatment with Gemcitabine 1000 mg/m2 and Cisplatin 25 mg/m2 on Days 1 and 8 of a 21 Day Cycle until tumor progression

SUMMARY:
The purpose of this study is to see if the investigational drug, RRx-001, an epigenetic agent, which turns on a number of beneficial genes that the tumor has silenced, can resensitize the tumor(s), in other words make it/them re-respond to gemcitabine and cisplatin, which, hopefully, will translate to a longer lifespan. The name of the open-label study, which means that patients will know what treatments they are receiving, is EPIC, a hybrid or combination of EPIgenetic for the mechanism of action of RRx-001 and Cholangiocarcinoma.

The study treatment is divided into two stages. During the first stage, patients will receive RRx-001, which is administered intravenously weekly, for a fixed time period of six weeks. At that time the second stage starts in which cisplatin and gemcitabine are reintroduced for as long as the tumors respond to them to determine whether resensitization has occurred.

The primary objective of this clinical trial is to evaluate the progression-free survival (PFS) of patients at 9 weeks after the reintroduction of gemcitabine and cisplatin.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of biliary tract adenocarcinoma/cholangiocarcinoma
* Must have locally advanced or distant metastatic disease that is not surgically curable
* Failed first-line chemotherapy
* Age ≥ 18 years
* Life expectancy of at least 12 weeks (3 months)
* Performance status 0 or 1
* Adequate liver, kidney, and bone marrow function

Exclusion Criteria:

* Symptomatic metastatic brain or meningeal tumors
* Investigational compound within 4 weeks of enrollment
* History of needing to permanently discontinue prior gemcitabine/ cisplatin regimen for reasons other than progression (i.e. toxicity)
* Any medical condition which, in the investigator's opinion, makes the patient unsuitable for participation
* Pregnant or nursing
* Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study or evaluation of the study results
* Albumin <2.8
* Uncontrolled or clinically relevant ascites
* Absolute contraindication for MRI imaging such as intracorporeal metal or pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-07-16 (Actual); Primary Completion 2016-05-10 (Actual); Study Completion 2016-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana De Jesus Acosta, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RRx-001 the Cisplatin and Gemcitabine
Started | 4
Completed | 3
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | RRx-001 the Cisplatin and Gemcitabine
Number analyzed (Participants) | 4
Age, Continuous [Median (Standard Deviation); unit: years] | 65.5 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Black or African American | 1
  White | 2
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Overall Objective Response (RECIST)
Description: Overall objective response (RECIST)
Time Frame: Baseline and every 6-8 weeks while on treatment until progression. Estimated 8 -24 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | RRx-001 the Cisplatin and Gemcitabine
Number analyzed (Participants) | 3
Participants | 3

ADVERSE EVENTS:
Arm/Group | RRx-001 the Cisplatin and Gemcitabine
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 2/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RRx-001 the Cisplatin and Gemcitabine (N=4)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RRx-001 the Cisplatin and Gemcitabine (N=4)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Renal Impairment (Renal and urinary disorders) | 1 (1)
Embolism (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No